CLINICAL TRIAL: NCT04074135
Title: Evaluation of the Natural History and Management of Von Hippel-Lindau (VHL) Associated Pancreatic Neuroendocrine Tumors
Brief Title: Natural History and Management of Von Hippel-Lindau (VHL) Associated Pancreatic Neuroendocrine Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 190135; 19-C-0135
Record Dates: First submitted 2019-08-28; First posted 2019-08-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01-08

CONDITIONS: VHL Pancreatic Neuroendocrine Tumors; Von Hippel-Lindau Disease; Neuroendocrine Tumors
Keywords: Pancreatic tumors; 68-Gallium DOTATATE; MEN1 syndrome; NETest; PNET
MeSH Terms: conditions — von Hippel-Lindau Disease; Neuroendocrine Tumors; Pancreatic Neoplasms; Multiple Endocrine Neoplasia Type 1; Neuroectodermal Tumors, Primitive | interventions — gallium Ga 68 dotatate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/ Arm 1 (Experimental): Study natural history of VHL pancreatic neuroendocrine tumors with yearly 68-Gallium DOTATATE PET/CT research scans.
  Interventions: Drug: 68-Gallium DOTATATE
- 2/ Arm 2 (No Intervention): Study natural history of VHL pancreatic neuroendocrine tumors without research scans.

INTERVENTIONS:
Drug: 68-Gallium DOTATATE — 68-Gallium DOTATATE, to be used in yearly PET/CT research scans
  Arms: 1/ Arm 1

SUMMARY:
Background:

People with von Hippel-Lindau (VHL) can have problems with a variety of organs, such as the pancreas. The disease can cause tumors of the pancreas. This can result in life-threatening complications. Researchers want to learn more about these pancreatic tumors and how to better detect them. This may help them design better future treatment and care for people with VHL disease.

Objective:

To better understand VHL disease that affects the pancreas and to test whether adding a certain type of scan (68-Gallium DOTATATE PET/CT) can further detect tumors.

Eligibility:

People ages 12 and older with VHL that causes tumors and cysts to grow in the pancreas

Design:

Participants will be screened with their medical records and imaging studies.

Participants will have an initial evaluation:

Participants will have their body examined by different doctors. This will depend on what types of symptoms they have.

Participants will have blood and urine tests

Participants will have images made of their body using one or more machines: They made have a CT or PET/CT scan in which they lie on a table that moves through a big ring. They may have an MRI in which they lie on a table that moves into a big tube. They may have an ultrasound that uses a small stick that produces sound waves to look at the body.

After the first visit, participants will be asked to return to the NIH. Some of the tests performed at the first visit will be repeated. Depending on their disease status, visits will be once a year or every 2 years for life.

DETAILED DESCRIPTION:
Background:

* Patients with the von Hippel-Lindau (VHL) familial cancer syndrome demonstrate manifestations in a variety of organs, including the pancreas. Pancreatic manifestations can range from benign cysts and micro cystic adenomas to neuroendocrine tumors of the pancreas which are capable of regional and distant metastases. These neuroendocrine tumors can result in life-threatening complications.
* This protocol is designed to identify VHL patients with pancreatic manifestations and to follow these patients with serial imaging studies, germ line genetic analysis, discovery of serum biomarkers, and novel imaging modalities such as 68-Gallium DOTATATE PET/CT scan.

Objective:

- To comprehensively and longitudinally evaluate the natural history of participants with VHL pancreatic neuroendocrine tumors and cystic lesions, estimating and defining their clinical spectrum.

Eligibility:

- Participants greater than or equal to 12 years of age diagnosed with VHL.

Design:

* Demographic data will be collected from the medical record and patient interview for each participant. Data will be securely stored in a computerized database.
* Participants will be evaluated by the urology, neurosurgery, brain oncology and/or ophthalmology personnel as indicated to rule out or manage other manifestations of VHL such as hemangioblastoma, renal cell cancer, and pheochromocytoma.
* Anatomical and functional clinical imaging studies, research blood and urine sample collection will be performed at each scheduled visit. Research 68-Gallium DOTATATE PET/CT imaging studies in adult participants will be performed, no more than once per year.
* Surgical resection of solid lesions of the pancreas will be recommended based on previously published criteria.
* Based on our analysis of likelihood of tumor growth or risk of metastasis, data will be analyzed every two years and appropriate revisions will be made to the surgical management guidelines, if indicated by data analysis.
* Up to 700 participants may receive the research 68-Gallium DOTATATE PET/CT imaging on this protocol.

ELIGIBILITY:
* INCLUSION CRITIERIA:

  1. Participants who have been diagnosed with VHL using the following criteria:

     -- Identification of a heterozygous germline pathogenic variant in VHL by molecular genetic testing.

     or

     -- Clinical criteria
  2. Participants with at least 1 pancreatic manifestation of VHL as documented on any non-invasive imaging study. These manifestations may include:

     * Pancreatic cyst(s)
     * Solid lesions suspicious for microcystic adenoma(s)
     * Solid enhancing lesions suspicious for PNET(s)
     * Any other solid lesion(s) of the pancreas
  3. Age greater than or equal to 12 years.
  4. Ability of participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Inability of participant to undergo serial non-invasive imaging.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 740 (Estimated)
Dates: Start 2020-06-02 (Actual); Primary Completion 2036-01-30 (Estimated); Study Completion 2036-07-01 (Estimated)

PRIMARY OUTCOMES:
Characterization of the natural and clinical histories of VHL pancreatic neuroendocrine tumors and cystic lesions | 15 years
  Characterization of the natural and clinical histories of VHL pancreatic neuroendocrine tumors and cystic lesions

SECONDARY OUTCOMES:
predictive value of 68-Gallium DOTATATE PET/CT imaging in patient population | at each scheduled visit
  mean uptake between these two groups of adult patients in which per patient uptake is defined as the average uptake of multiple lesions detected in each patient
growth rate in solid pancreatic tumors | at each scheduled visit
  graded tumor biopsy
distribution of time from initial presentation with pancreatic tumors to the time that surgery is recommended | at each scheduled visit, until surgery is recommended
  median amount of time from initial presentation with pancreatic tumors to the time that surgery is recommended

CONTACTS AND LOCATIONS:
Overall Officials: Naris Nilubol, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-C-0135.html